CLINICAL TRIAL: NCT05583279
Title: Implementation of Dialectical Behavioral Therapy in Juvenile Justice to Reduce Self-Harm and Increase Quality of Life: A Pilot Test
Brief Title: Dialectical Behavioral Therapy in Juvenile Justice
Acronym: DBT-A&JJS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We never started the study.
Sponsor: The Catholic University of America (Other)
Collaborators: Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CUA-002
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Non-Suicidal Self Injury; Suicide; Self-harm; Emotion Regulation
Keywords: dialectical behavioral therapy; adolescents; self-injury; suicide; juvenile justice
MeSH Terms: conditions — Self-Injurious Behavior; Suicide; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: The proposed project consists of a mixed-methods cross-over design involving a three-phase clinical trial aimed at assessing the feasibility, acceptability, and preliminary effectiveness of comprehensive DBT-A adapted for youth in the GAJJS. DBT-A/outcomes will be assessed across two different levels of care (i.e., at short- vs. long-term facilities) and service delivery methods (i.e., in-person vs. telehealth).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 2 (Experimental): Cohort 1 and 2 youth will then complete baseline assessments (see 4.5) and Cohort 2 will continue receiving TAU while Cohort 1 begins receiving DBT-A (randomized by facility to either in-person or via telehealth delivery) for the next six months while Cohort 1 staff continue consultation with DBT-A. After six months, Phase 2 of this study will conclude with the youth of Cohorts 1 and 2 completing their first follow-up assessment. The implementation plan will be altered accordingly based on feedback from stakeholders prior to the start of Phase 2. The modified implementation plan will be used in the training of the staff in DBT-A at the second four facilities prior to the launch of Phase 3.
  Interventions: Behavioral: Dialetical Behavioral Therapy for Adolescents
- No intervention (Active Comparator): Cohort 2 will not receive any treatment during Phase 2 of the study, which is the first part of the clinical trial. They will serve as a comparison group for Cohort 1.
  Interventions: Behavioral: Dialetical Behavioral Therapy for Adolescents
- Phase 3 (Active Comparator): Phase 3 will begin with making any modifications to the treatment protocol based on a review of feedback from stakeholder interviews from Phase 2. Cohort 2 facilities will be randomized to delivering DBT-A in-person or via telehealth (one long-term and one short-term facility will be assigned to each condition). Staff in Cohort 2 will receive training and consultation in DBT-A and implement either telehealth or in-person delivered DBT-A in their facilities. Cohort 1 facilities will cross-over from in-person delivery of DBT-A to telehealth delivery, or vice-versa, thereby facilitating a within-facility comparison of DBT-A delivery methods. After six months, Phase 3 will conclude with the youth of Cohorts 1 and 2 completing their second follow-up assessment and all stakeholders of Cohorts 1 and 2 completing stakeholder interviews.
  Interventions: Behavioral: Dialetical Behavioral Therapy for Adolescents

INTERVENTIONS:
Behavioral: Dialetical Behavioral Therapy for Adolescents — DBT is an evidence-based treatment for individuals with complex clinical presentations, including borderline personality disorder (BPD), suicidality, and NSSI. Standard DBT (which includes individual therapy, skills group, between-session skills coaching, and peer consultation for therapists) is associated with symptom reductions in patients across a variety of domains, including BPD symptoms, SA, NSSI, hospitalizations, and social functioning. DBT focuses on teaching skills (e.g., emotion regulation) and facilitating the replacement of impulsive and/or ineffective behaviors (e.g., NSSI), with more effective/skillful behaviors.

SUMMARY:
Self-injurious thoughts and behaviors (SITBs) are a serious public health concern, particularly for youth involved in the juvenile justice system (JJS), which the Georgia State Juvenile Justice System (GAJJS) intends to address by the implementation of Dialectical Behavior Therapy (DBT) in its JJS facilities. This proposal aims to support and study the GAJJS' pilot implementation of DBT at its facilities using a mixed-methods cross-over design involving a three-phase clinical trial assessing the feasibility, acceptability, and preliminary effectiveness of DBT-A adapted for youth in the GAJJS. By the end of the proposed project, the investigators will have (1) established a research team to continue researching SITB interventions in the GAJJS, (2) developed protocols for implementing and evaluating DBT-A adapted for the JJS delivered in person and via telehealth, and (3) preliminary data on the feasibility, acceptability, and effectiveness of DBT-A adapted for the JJS.

DETAILED DESCRIPTION:
Self-injurious thoughts and behaviors (SITBs) are a serious public health concern across the United States, and youth involved in the juvenile justice system (JJS) are at particularly high-risk for SITBs. As part of the Georgia State Juvenile Justice System (GAJJS)'s decades long collaboration with researchers to reduce the rates of suicide and non-suicidal self-injury (NSSI) among youth under their care, they identified Dialectical Behavior Therapy (DBT) as an ideal intervention to fit their needs and subsequently made plans to pilot an adapted DBT for JJS in a portion of their facilities. DBT is an evidence-based treatment for individuals with complex clinical presentations, which has demonstrated effectiveness at reducing SITBs when adapted for adolescents (DBT-A). Despite its adoption by several JJSs, the effectiveness of DBT-A has yet to be empirically evaluated. A controlled evaluation of DBT-A in JJS is desperately needed to develop a framework for implementation and assess its feasibility, acceptability, and preliminary effectiveness. However, GAJJS does not have the resources or expertise to evaluate the intervention's feasibility, acceptability, and preliminary effectiveness on their own. Therefore, this project proposes to capitalize on this unique opportunity to investigate the GAJJS's implementation of DBT across eight pilot facilities. The investigators propose a mixed-methods cross-over design involving a three-phase clinical trial aimed at assessing the feasibility, acceptability, and preliminary effectiveness of DBT-A adapted for youth in the GAJJS. SITB-related outcomes and DBT-A's feasibility and acceptability will be assessed across two different levels of care (i.e., at short- vs. long-term facilities) and service delivery methods (i.e., in-person vs. telehealth). The project will use feedback from stakeholders, collected at multiple timepoints, to design and iterate the adapted DBT-A program to maximize its feasibility, acceptability, and effectiveness in the GAJJS. The clinical trial will use administrative clinical, health, and educational data of JJS-involved youth to assess how effective DBT-A is at reducing self-harming behaviors and associated risk factors (i.e., deficits in distress tolerance, emotion dysregulation, and interpersonal skills). By the end of the proposed project, the investigators will have (1) established a research team to continue researching SITB interventions in the GAJJS; (2) developed protocols for implementing and evaluating DBT-A adapted for the JJS delivered in person and via telehealth; and (3) preliminary data on the feasibility, acceptability, and effectiveness of DBT-A adapted for the JJS. The investigators will then have the personnel, intervention, and preliminary data to submit an R01 to evaluate the effectiveness of our JJS-adapted DBT-A in a fully powered randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* must be in the custody of the GAJJS and placed at one of the eight facilities participating in the study,
* can speak, read, and understand English well enough to participate in a DBT-A therapy program,
* there is written informed assent, and
* verbal parental/guardian or youth advocate informed consent has been obtained.

Exclusion Criteria:

- any youth who are cognitively/decisionally impaired, the GAJJS conducts detailed psycho-diagnostic evaluations on all youth during their intake evaluation - and, part of this evaluation includes a thorough mental status exam, conducted by one of the mental health staff.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The short form of the self-injurious thoughts and behaviors interview (SITBI) | six months to 12 months for cohort 1, six months for cohort 2
  Measures changes in suicidal and non-suicidal self-injurious thoughts and behaviors
The Life Problems Inventory (LPI) | six months to 12 months for cohort 1, six months for cohort 2
  Measures the four core treatment components of DBT-A: emotion dysregulation, impulsivity, interpersonal chaos, and confusion about self.
The DBT-Ways of Coping Check List (DBT-WCCL) | six months to 12 months for cohort 1, six months for cohort 2
  Measures the use of DBT skills and dysfunctional, non-DBT coping strategies
The Acceptance and Action Questionnaire II (AAQ-II) | six months to 12 months for cohort 1, six months for cohort 2
  a self-report measure of experiential avoidance

CONTACTS AND LOCATIONS:
Overall Officials: Melissa D Grady, PhD, Principal Investigator — Catholic University
Locations (1):
- Catholic University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
The Catholic University of America is committed to the open and timely dissemination of research outcomes. Investigators in this proposed program recognize that promising new methods, technologies, data, software programs, and insights may arise during the course of their research. All investigators are aware of and agree to abide by the principles for sharing research resources, as described by NIH in, "Principles and Guidelines for Recipients of NIH Research Grants and Contracts on Obtaining and Disseminating Biomedical Research Programs".
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: the data will become available one year after completion of the trial and will be available for three years.
Access Criteria: Researchers who work within juvenile justice systems.

REFERENCES:
- [Background] Ludtke J, In-Albon T, Schmeck K, Plener PL, Fegert JM, Schmid M. Nonsuicidal Self-Injury in Adolescents Placed in Youth Welfare and Juvenile Justice Group Homes: Associations with Mental Disorders and Suicidality. J Abnorm Child Psychol. 2018 Feb;46(2):343-354. doi: 10.1007/s10802-017-0291-8. PMID 28374220
- [Background] Abram KM, Choe JY, Washburn JJ, Teplin LA, King DC, Dulcan MK. Suicidal ideation and behaviors among youths in juvenile detention. J Am Acad Child Adolesc Psychiatry. 2008 Mar;47(3):291-300. doi: 10.1097/CHI.0b013e318160b3ce. PMID 18216737
- [Background] Linehan MM. Dialectical behavior therapy for borderline personality disorder. Theory and method. Bull Menninger Clin. 1987 May;51(3):261-76. No abstract available. PMID 3580661
- [Background] Kothgassner OD, Goreis A, Robinson K, Huscsava MM, Schmahl C, Plener PL. Efficacy of dialectical behavior therapy for adolescent self-harm and suicidal ideation: a systematic review and meta-analysis. Psychol Med. 2021 May;51(7):1057-1067. doi: 10.1017/S0033291721001355. Epub 2021 Apr 20. PMID 33875025
- [Background] Moscicki EK. Gender differences in completed and attempted suicides. Ann Epidemiol. 1994 Mar;4(2):152-8. doi: 10.1016/1047-2797(94)90062-0. PMID 8205283
- [Background] Clarke S, Allerhand LA, Berk MS. Recent advances in understanding and managing self-harm in adolescents. F1000Res. 2019 Oct 24;8:F1000 Faculty Rev-1794. doi: 10.12688/f1000research.19868.1. eCollection 2019. PMID 31681470
- [Background] Cibis A, Mergl R, Bramesfeld A, Althaus D, Niklewski G, Schmidtke A, Hegerl U. Preference of lethal methods is not the only cause for higher suicide rates in males. J Affect Disord. 2012 Jan;136(1-2):9-16. doi: 10.1016/j.jad.2011.08.032. Epub 2011 Sep 19. PMID 21937122
- [Background] Carmel A, Rose ML, Fruzzetti AE. Barriers and solutions to implementing dialectical behavior therapy in a public behavioral health system. Adm Policy Ment Health. 2014 Sep;41(5):608-14. doi: 10.1007/s10488-013-0504-6. PMID 23754686
- [Background] Thorpe KE, Zwarenstein M, Oxman AD, Treweek S, Furberg CD, Altman DG, Tunis S, Bergel E, Harvey I, Magid DJ, Chalkidou K. A pragmatic-explanatory continuum indicator summary (PRECIS): a tool to help trial designers. J Clin Epidemiol. 2009 May;62(5):464-75. doi: 10.1016/j.jclinepi.2008.12.011. PMID 19348971
- [Background] Ruch DA, Sheftall AH, Schlagbaum P, Fontanella CA, Campo JV, Bridge JA. Characteristics and Precipitating Circumstances of Suicide Among Incarcerated Youth. J Am Acad Child Adolesc Psychiatry. 2019 May;58(5):514-524.e1. doi: 10.1016/j.jaac.2018.07.911. Epub 2019 Jan 23. PMID 30768395
- [Background] Wilkinson PO. Dialectical Behavior Therapy-A Highly Effective Treatment for Some Adolescents Who Self-harm. JAMA Psychiatry. 2018 Aug 1;75(8):786-787. doi: 10.1001/jamapsychiatry.2018.1079. No abstract available. PMID 29926089
- [Background] James AC, Taylor A, Winmill L, Alfoadari K. A Preliminary Community Study of Dialectical Behaviour Therapy (DBT) with Adolescent Females Demonstrating Persistent, Deliberate Self-Harm (DSH). Child Adolesc Ment Health. 2008 Sep;13(3):148-152. doi: 10.1111/j.1475-3588.2007.00470.x. Epub 2007 Dec 14. PMID 32847177
- [Background] McAllister-Williams RH, Young AH. Pindolol augmentation of antidepressant therapy. Br J Psychiatry. 1998 Dec;173:536-7. doi: 10.1192/bjp.173.6.536b. No abstract available. PMID 9926087
- [Background] DeCou CR, Comtois KA, Landes SJ. Dialectical Behavior Therapy Is Effective for the Treatment of Suicidal Behavior: A Meta-Analysis. Behav Ther. 2019 Jan;50(1):60-72. doi: 10.1016/j.beth.2018.03.009. Epub 2018 Mar 22. PMID 30661567
- [Background] Lynch TR, Chapman AL, Rosenthal MZ, Kuo JR, Linehan MM. Mechanisms of change in dialectical behavior therapy: theoretical and empirical observations. J Clin Psychol. 2006 Apr;62(4):459-80. doi: 10.1002/jclp.20243. PMID 16470714
- [Background] Rathus JH, Miller AL. Dialectical behavior therapy adapted for suicidal adolescents. Suicide Life Threat Behav. 2002 Summer;32(2):146-57. doi: 10.1521/suli.32.2.146.24399. PMID 12079031
- [Background] Carson-Wong A, Hughes CD, Rizvi SL. The effect of therapist use of validation strategies on change in client emotion in individual dbt treatment sessions. Personal Disord. 2018 Mar;9(2):165-171. doi: 10.1037/per0000229. Epub 2016 Dec 5. PMID 27918168
- [Background] Cooperman NA, Rizvi SL, Hughes CD, Williams JM. Field Test of a Dialectical Behavior Therapy Skills Training-Based Intervention for Smoking Cessation and Opioid Relapse Prevention in Methadone Treatment. J Dual Diagn. 2019 Jan-Mar;15(1):67-73. doi: 10.1080/15504263.2018.1548719. Epub 2019 Jan 15. PMID 30646819
- [Background] Rizvi SL, Hughes CD, Hittman AD, Vieira Oliveira P. Can Trainees Effectively Deliver Dialectical Behavior Therapy for Individuals With Borderline Personality Disorder? Outcomes From a Training Clinic. J Clin Psychol. 2017 Dec;73(12):1599-1611. doi: 10.1002/jclp.22467. Epub 2017 Feb 21. PMID 28221671
- [Background] Pistorello J, Jobes DA, Compton SN, Locey NS, Walloch JC, Gallop R, Au JS, Noose SK, Young M, Johnson J, Dickens Y, Chatham P, Jeffcoat T, Dalto G, Goswami S. Developing Adaptive Treatment Strategies to Address Suicidal Risk in College Students: A Pilot Sequential, Multiple Assignment, Randomized Trial (SMART). Arch Suicide Res. 2017 Oct-Dec;22(4):644-664. doi: 10.1080/13811118.2017.1392915. Epub 2018 Feb 12. PMID 29220633
- [Background] Andreasson K, Krogh J, Rosenbaum B, Gluud C, Jobes DA, Nordentoft M. The DiaS trial: dialectical behavior therapy versus collaborative assessment and management of suicidality on self-harm in patients with a recent suicide attempt and borderline personality disorder traits - study protocol for a randomized controlled trial. Trials. 2014 May 29;15:194. doi: 10.1186/1745-6215-15-194. PMID 24885904
- [Background] David Rudd M, Bryan CJ, Jobes DA, Feuerstein S, Conley D. A Standard Protocol for the Clinical Management of Suicidal Thoughts and Behavior: Implications for the Suicide Prevention Narrative. Front Psychiatry. 2022 Jul 12;13:929305. doi: 10.3389/fpsyt.2022.929305. eCollection 2022. PMID 35903634
- [Background] Jobes DA, Chalker SA. One Size Does Not Fit All: A Comprehensive Clinical Approach to Reducing Suicidal Ideation, Attempts, and Deaths. Int J Environ Res Public Health. 2019 Sep 26;16(19):3606. doi: 10.3390/ijerph16193606. PMID 31561488
- [Background] Maclure M, Mittleman MA. Should we use a case-crossover design? Annu Rev Public Health. 2000;21:193-221. doi: 10.1146/annurev.publhealth.21.1.193. PMID 10884952
- [Background] Chugani CD, Mitchell ME, Botanov Y, Linehan MM. Development and Initial Evaluation of the Psychometric Properties of the Dialectical Behavior Therapy Barriers to Implementation Scale (BTI-S). J Clin Psychol. 2017 Dec;73(12):1704-1716. doi: 10.1002/jclp.22478. Epub 2017 Apr 5. PMID 28380249
- [Background] Aarons GA. Mental health provider attitudes toward adoption of evidence-based practice: the Evidence-Based Practice Attitude Scale (EBPAS). Ment Health Serv Res. 2004 Jun;6(2):61-74. doi: 10.1023/b:mhsr.0000024351.12294.65. PMID 15224451
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Dimeff LA, Woodcock EA, Harned MS, Beadnell B. Can dialectical behavior therapy be learned in highly structured learning environments? Results from a randomized controlled dissemination trial. Behav Ther. 2011 Jun;42(2):263-75. doi: 10.1016/j.beth.2010.06.004. Epub 2011 Jan 26. PMID 21496511
- [Background] Fox KR, Harris JA, Wang SB, Millner AJ, Deming CA, Nock MK. Self-Injurious Thoughts and Behaviors Interview-Revised: Development, reliability, and validity. Psychol Assess. 2020 Jul;32(7):677-689. doi: 10.1037/pas0000819. Epub 2020 Apr 23. PMID 32324021
- [Background] Nock MK, Holmberg EB, Photos VI, Michel BD. Self-Injurious Thoughts and Behaviors Interview: development, reliability, and validity in an adolescent sample. Psychol Assess. 2007 Sep;19(3):309-17. doi: 10.1037/1040-3590.19.3.309. PMID 17845122
- [Background] Neacsiu AD, Rizvi SL, Linehan MM. Dialectical behavior therapy skills use as a mediator and outcome of treatment for borderline personality disorder. Behav Res Ther. 2010 Sep;48(9):832-9. doi: 10.1016/j.brat.2010.05.017. Epub 2010 May 23. PMID 20579633
- [Background] Harned MS, Korslund KE, Schmidt SC, Gallop RJ. The Dialectical Behavior Therapy Adherence Coding Scale (DBT ACS): Psychometric properties. Psychol Assess. 2021 Jun;33(6):552-561. doi: 10.1037/pas0000999. Epub 2021 Mar 25. PMID 33764118
- See also: Center for Disease Control Injury Data — https://www.cdc.gov/injury/wisqars/index.html
- See also: Ford JD, Chapman JF, Hawke J, Albert D. Trauma among youth in the juvenile justice system: Critical issues and new directions. National Center for Mental Health and Juvenile Justice. 2007;6:2007. — https://www.courts.ca.gov/documents/BTB25-1G-02.pdf
- See also: Wilks CR, Gurtovenko K. Virtual delivery of dialectical behavior therapy. In: Rolnik A, ed. Advances in online therapy. ; in press. — https://bpded.biomedcentral.com/articles/10.1186/s40479-021-00167-5
- See also: National Action Alliance for Suicide Prevention: Research Prioritization Task Force. A prioritized research agenda for suicide prevention: An action plan to save lives. . 2014. — https://theactionalliance.org/resource/prioritized-research-agenda-suicide-prevention-action-plan-save-lives
- See also: Courtney-Seidler, E. A., Burns, K., Zilber, I., & Miller, A. L. (2014). Adolescent suicide and self-injury: Deepening the understanding of the biosocial theory and applying dialectical behavior therapy. — https://www.semanticscholar.org/paper/Adolescent-suicide-and-self-injury%3A-Deepening-the-Courtney-Seidler-Burns/5a85298db525d7103beb74b49a44066d47f10d95
- See also: Drake EK, Barnoski RP. Recidivism findings for the juvenile rehabilitation administration's mentoring program. Washington State Institute for Public Policy; 2006. — https://www.wsipp.wa.gov/ReportFile/947/Wsipp_Recidivism-Findings-for-the-Juvenile-Rehabilitation-Administrations-Mentoring-Program-Final-Report_Full-Report.pdf
- See also: Harned MS, Coyle TN, Garcia NM. The inclusion of ethnoracial, sexual, and gender minority groups in randomized controlled trials of dialectical behavior therapy: A systematic review of the literature. Clinical Psychology: Science and Practice. 2022. — https://www.apa.org/pubs/journals/cps
- See also: BOND DM, HOMAN J, BEACH B. DBT in juvenile justice programs. Dialectical Behavior Therapy in Clinical Practice: Applications across Disorders and Settings. 2020;159. — https://www.guilford.com/books/Dialectical-Behavior-Therapy-in-Clinical-Practice/Dimeff-Rizvi-Koerner/9781462544622
- See also: Schatten TH, Hughes CD. The patient with nonsuicidal self-injury. — https://www.amazon.com/Inpatient-Psychiatric-Nursing-2nd-Interventions/dp/0826135439
- See also: Hughes CD, Rizvi SL. Applying a cognitive-behavioral, principle-based approach to the treatment of personality disorders: An extension of Rosenthal, Wyatt, and McMahon. — https://www.cambridge.org/core/books/abs/cambridge-handbook-of-personality-disorders/treatment/888E924B72635427D8E91B4733AAC796
- See also: Hughes CD, King AM, Kranzler A, et al. Anxious and overwhelming affects and repetitive negative thinking as ecological predictors of self-injurious thoughts and behaviors. Cognitive Therapy and Research. 2019;43(1):88-101. — https://einstein.pure.elsevier.com/en/publications/anxious-and-overwhelming-affects-and-repetitive-negative-thinking
- See also: Guarino D, Lesnewich LM, Clemow L, Hughes CD, Rizvi SL. Implementing a dbt group intervention in a primary care setting: A feasibility and acceptability study. . 2020;54:S333. — https://rucore.libraries.rutgers.edu/rutgers-lib/64610/
- See also: Jobes DA. Commonsense recommendations for standard care of suicidal risk. Journal of Health Service Psychology. 2020;46(4):155-163. — https://link.springer.com/article/10.1007/s42843-020-00020-3
- See also: Miller AL, Rathus JH, Linehan MM. Dialectical behavior therapy with suicidal adolescents. Guilford Press; 2006. — https://www.guilford.com/books/Dialectical-Behavior-Therapy-with-Suicidal-Adolescents/Miller-Rathus-Linehan/9781462532056
- See also: Rathus JH, Miller AL. DBT skills manual for adolescents. Guilford Publications; 2014. — https://www.guilford.com/books/DBT-Skills-Manual-for-Adolescents/Rathus-Miller/9781462515356
- See also: Ford JD. TARGET: Trauma affect regulation: Guide for education and therapy. University of Connecticut Health Center. 2006. — https://www.cttntraumatraining.org/uploads/4/6/2/3/46231093/target.pdf
- See also: Rathus JH, Wagner D, Miller AL. Psychometric evaluation of the life problems inventory, a measure of borderline personality features in adolescents. Journal of Psychology & Psychotherapy. 2015;5(4):1-9. — https://www.longdom.org/open-access/psychometric-evaluation-of-the-life-problems-inventory-a-measure-of-borderline-personality-features-in-adolescents-2161-0487-1000198.pdf
- See also: Harned MS, Schmidt SC, Korslund KE. No title. The dialectical behavior therapy adherence checklist for individual therapy (DBT AC-I). 2021. — https://static1.squarespace.com/static/610d7fa3dbc3322bc501ff8e/t/616f62830e9797618438160c/1634689668247/DBT+AC-I+Training+Manual+v1.0.pdf
- See also: Attkisson CC, Greenfield TK. The client satisfaction questionnaire (CSQ) scales and the service satisfaction scale-30 (SSS-30). Outcomes assessment in clinical practice. 1996;120(7):120-127. — http://apntoolkit.mcmaster.ca/index.php?view=article&id=94%3Aclient-satisfaction-questionnaire-csq-8&format=pdf&option=com_content